CLINICAL TRIAL: NCT02739178
Title: The Sukhshanti Study: a Controlled Before-and-after Mixed Methods Study of the Effect of a Sanitation Intervention on Women's Health in Bihar, India
Brief Title: The Sukhshanti Study: Effect of a Sanitation Intervention on Women's Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively inactivated by IRB due to no response for Continuing Review
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6580 Norman
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSF Sanitation intervention (Experimental): This arm will receive the GSF sanitation intervention, a community-level sanitation intervention
  Interventions: Other: GSF Intervention
- Comparator (No Intervention): This arm will receive the GSF intervention in 2017 or later.

INTERVENTIONS:
Other: GSF Intervention — Intervention utilizes community-based demand generation matched with supply side improvements to improve access and use of sanitation facilities in rural communities. This is complimented with multi-stakeholder engagement to promote cooperation and coordination with national, state, and local stakeholders.
  Arms: GSF Sanitation intervention

SUMMARY:
The study will measure the impact of sanitation access on women and girl's social and emotional health, behaviors, and quality of life in rural India before and after a sanitation intervention compared to a comparison group that will receive the same intervention at a later date.

DETAILED DESCRIPTION:
This mixed-methods, quasi-experimental study will evaluate the extent to which the Global Sanitation Fund (GSF) sanitation program in Bihar, India improves health and well-being among women and girls. Our study consists of a controlled before-and-after (CBA) study with an embedded ethnography.

Specific objectives are:

* Measure the effect of the GSF intervention on sanitation-related psychosocial stress (SRPS), generalized psychosocial stress (PSS), perceived quality of life, hair cortisol, and urogenital health among women between the ages of 14 and 65.
* Measure changes in sanitation adoption (e.g.: sanitation access and exclusive use) among individuals / households receiving the GSF intervention.
* Document individual and community experiences with sanitation, intervention participation, and latrine coverage through ethnographic methods.

ELIGIBILITY:
Inclusion Criteria:

* between 14 years to 65 years old
* live in geographic area receiving GSF sanitation intervention in 2016
* live in geographic areas matched to intervention communities

Exclusion Criteria:

* less than 25 years old and not reached menarche
* greater than 25 years old and never married
* refusal to participate

Ages: 14 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1275 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Sanitation-Related Psychosocial Stress Scale (SRPS) | 12 month follow-up
  The SRPS consist of 25 yes/no questions on experiences related to sanitation within the past thirty days of the date the SRPS is completed.This SRPS Scale specifically includes questions related to defecation, menstrual hygiene management, and post-defecation cleaning - the three behaviors that have the greatest contribution to sanitation-related psychosocial stress among women in India.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS10) | 12 month follow-up
  A measure for non-specific perceived stress. The PSS10 is the short form of the PSS and consist of 10 items rated on a 5-point Likert scale (0 to 4). Scores are calculated by reverse scoring items with positive wording and summing across all items for a final score of 0 to 40. The PSS10 is not a diagnostic scale.
Kessler Psychological Distress Scale (K10) | 12 month follow-up
  The K10 provides a measure of non-specific psychological distress and consists of 10 items rated on a 5-point Likert scale (1 to 5). Scores are calculated by summing response across each item.
The WHO5 Well-Being Index (WHO-5) | 12 month follow-up
  The WHO5 consist of 5 items rated on a 6-point Likert scale (0 to 5) related to subjective well-being, vitality, and mood.
Self-reported urogenital infections | 12 month follow-up
  Urogenital infections, a health outcome linked to both menstrual hygiene management practices and sanitation access (Das et al., 2015) will be identified through self-report of any one of the following four symptoms: abnormal vaginal discharge (unusual texture / color and/or more abundant discharge than normal), burning or itching of the genitalia, burning or itching when urinating, or having genital sores.
Hair cortisol | 12 month follow-up
  Hair cortisol will be assessed in a sub-sample of women in both intervention and comparison communities.
Sleep duration | 12 month follow-up
  Sleep duration will be assessed through a variety of self-report methods. The investigators will adapt questions from the Pittsburgh Sleep Quality Index that assess sleep duration over the past month: 1. During this past month, how many hours of actual sleep did the participant usually get at night? (Herring et al., 2013). The investigators will also ask the following questions: 1. To the best of the participant's knowledge, what time did the participant go to bed last night? 2. To the best of the participant's knowledge, what time did the participant wake up this morning?

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Cumming, Mr., Study Director — London School of Hygiene and Tropical Medicine; Kathleen O'Reilly, PhD, Study Director — Texas A&M University; Seema Kulkarni, Study Director — Society for the Promotion of Participatory Ecosystem Management (SOPPECOM); Robert Dreibelbis, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- NEERMAN, Mumbai, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available after completion of the study.